CLINICAL TRIAL: NCT00377949
Title: The Natural History and Outcome of Patients With Scleroderma at High Risk for or With Early Pulmonary Hypertension
Brief Title: Multi-center, Web Based Observational Study of Pulmonary Hypertension in Scleroderma Patients
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Virginia Steen, MD, Project Principal Investigator, Georgetown University
Other Study IDs: IRB # 04-227
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Systemic Sclerosis; Scleroderma; Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: Systemic Sclerosis; Scleroderma; Pulmonary Hypertension; PHAROS; PHROS; Exercise Echocardiogram; Pulmonary Functional Tests; Six minute walk tests; 6 minute walk tests; Right heart catheterization
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum stored for future analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the timeline of progression from pre-pulmonary hypertension to diagnosable pulmonary hypertension based on right heart catheterization. Moreover, to determine the timeline for progression from diagnosable pulmonary hypertension to clinical worsening of disease as defined as death, hospitalization, or worsening of PHT symptoms.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare, often fatal idiopathic disease, which has no effective therapy. One of the most major complications of systematic sclerosis is pulmonary hypertension (PHT), which is now the cause of all scleroderma related deaths. New therapeutic advances have improved short-term management of pulmonary hypertension in scleroderma, but long-term outcomes are unknown. With this in mind, Dr. Steen has developed Pulmonary Hypertension Assessment Registry of Scleroderma (PHAROS), a preventive, multi-center, web based observational study that looks at the natural history and outcome of scleroderma patients who are at high risk or have early pulmonary hypertension. Patients entered into the registry will be followed in prospective fashion noting the clinical course of disease by both scheduled and event driven follow up. A thorough baseline history will be collected to determine key prognostic and correlative factors for both disease prevalence and progression. Yearly follow up consisting of questionnaires, pulmonary function tests, echocardiogram, 6 minute walk tests and predefined patient characteristics will also be conducted to further understand and note the progression of scleroderma related PAH. Event driven follow up will occur to record findings and record specific predetermined events in the clinical course of disease.

ELIGIBILITY:
1. Global Inclusion Criteria

   * Eligible patients must meet all of the following inclusion criteria:
   * Patient ≥ 18 years with a clinical diagnosis of SSc (ACR criteria or the LeRoy criteria for limited or diffuse scleroderma
2. Specific Inclusion Criteria

   * Diagnosis of "pre" pulmonary arterial hypertension defined as:
   * Echocardiogram with a resting sPAP of ≥ 40mmHg Or
   * Pulmonary function test with FVC >70% and a DLCO <55% of predicted or a FVC/DLco ratio >1.6. or
   * Right heart catheterization which shows or a mean PA pressure > 30mmHg with exercise (with a mPAP < 25mmHg at rest)

Patients entered as a 'pre'-pulmonary arterial hypertension who then undergo right heart catheterization and are found to have pulmonary arterial hypertension, pulmonary venous hypertension or diastolic dysfunction or pulmonary hypertension secondary to interstitial lung disease will be followed as a definite PH patient and classified into the appropriate category.

* Diagnosis of definite pulmonary hypertension Patients with pulmonary hypertension with a right heart catheterization showing a mean PA pressure > 25mmHg, diagnosed in the past 6 months.

Classification of PH Group 1 PAH - Patients with mPAP ≥ 25mmHg with a wedge < 15mmHg Group 2 PVH - Patients who have a mean PA pressure ≥ 25mmHg with a wedge pressure which is > 15 mmHg Group 3 PH-ILD Patients who have a mean PA pressure ≥ 25mmHg (on right heart catheterization) who have moderate to severe interstitial fibrosis on HRCT scan with a FVC and TLC < 65% predicted

b. Exclusion Criteria

* Diagnosis and treatment of pulmonary hypertension for > 6 months
* Patients with known severe interstitial fibrosis, pulmonary thrombotic disease, heart failure, cardiomyopathy,history of coronary artery disease or other cardio-pulmonary problems which could cause pulmonary hypertension are not eligible for the 'pre'-pulmonary hypertension but do qualify for the definite pulmonary hypertension group if they have a right heart catheterization showing a mean PAH >25mmHg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care, rheumatology and pulmonary hypertension clinics.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2005-02; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Hypertension Progression | 10 years
  The primary objective of the study is to determine the timeline of progression from pre-pulmonary hypertension to diagnosable pulmonary hypertension based on right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Virginia D. Steen, MD, Principal Investigator — Georgetown University
Locations (25):
- United States (25):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - John Hopkins University Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical School, Boston, Massachusetts
  - University of Massachussetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan-Scleroderma Program, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Center for Rheumatology, Albany, New York
  - North Shore Long Island Jewish Medical Center, New Hyde Park, New York
  - Hospital for Special Surgery, New York, New York
  - Cornell University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Young RH, Mark GJ. Pulmonary vascular changes in scleroderma. Am J Med. 1978 Jun;64(6):998-1004. doi: 10.1016/0002-9343(78)90455-2. PMID 148843
- [Background] Salerni R, Rodnan GP, Leon DF, Shaver JA. Pulmonary hypertension in the CREST syndrome variant of progressive systemic sclerosis (scleroderma). Ann Intern Med. 1977 Apr;86(4):394-9. doi: 10.7326/0003-4819-86-4-394. PMID 848800
- [Background] Stupi AM, Steen VD, Owens GR, Barnes EL, Rodnan GP, Medsger TA Jr. Pulmonary hypertension in the CREST syndrome variant of systemic sclerosis. Arthritis Rheum. 1986 Apr;29(4):515-24. doi: 10.1002/art.1780290409. PMID 3707629
- [Background] Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, Groves BM, Tapson VF, Bourge RC, Brundage BH, Koerner SK, Langleben D, Keller CA, Murali S, Uretsky BF, Clayton LM, Jobsis MM, Blackburn SD, Shortino D, Crow JW; Primary Pulmonary Hypertension Study Group. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1996 Feb 1;334(5):296-301. doi: 10.1056/NEJM199602013340504. PMID 8532025
- [Background] Steen VD, Ziegler GL, Rodnan GP, Medsger TA Jr. Clinical and laboratory associations of anticentromere antibody in patients with progressive systemic sclerosis. Arthritis Rheum. 1984 Feb;27(2):125-31. doi: 10.1002/art.1780270202. PMID 6607734
- [Background] Murata I, Takenaka K, Yoshinoya S, Kikuchi K, Kiuchi T, Tanigawa T, Ito K. Clinical evaluation of pulmonary hypertension in systemic sclerosis and related disorders. A Doppler echocardiographic study of 135 Japanese patients. Chest. 1997 Jan;111(1):36-43. doi: 10.1378/chest.111.1.36. PMID 8995990
- [Background] Denton CP, Cailes JB, Phillips GD, Wells AU, Black CM, Bois RM. Comparison of Doppler echocardiography and right heart catheterization to assess pulmonary hypertension in systemic sclerosis. Br J Rheumatol. 1997 Feb;36(2):239-43. doi: 10.1093/rheumatology/36.2.239. PMID 9133938
- [Background] MacGregor AJ, Canavan R, Knight C, Denton CP, Davar J, Coghlan J, Black CM. Pulmonary hypertension in systemic sclerosis: risk factors for progression and consequences for survival. Rheumatology (Oxford). 2001 Apr;40(4):453-9. doi: 10.1093/rheumatology/40.4.453. PMID 11312386
- [Background] Yousem SA. The pulmonary pathologic manifestations of the CREST syndrome. Hum Pathol. 1990 May;21(5):467-74. doi: 10.1016/0046-8177(90)90002-m. PMID 2186993